CLINICAL TRIAL: NCT02930668
Title: Double-blind, Randomised, Placebo-controlled Study to Evaluate Benefit of Glucosanol™ in Reducing Body Weight in Overweight and Moderately Obese Subjects
Brief Title: Efficacy and Safety of Glucosanol™ in Body Weight Reduction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: InQpharm Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: INQ/024115
Record Dates: First submitted 2016-10-10; First posted 2016-10-12 (Estimated); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): The placebo is identical in shape, colour and size to the active comparator with the active ingredient replaced with microcrystalline cellulose.
  Subjects will take 2 capsules three times a day, 30 mins before meals.
  Interventions: Dietary Supplement: Placebo
- Low dose (Glucosanol 350mg) (Experimental): Each capsule contains Glucosanol / Phaselite 350mg
  Subjects will take 2 capsules three times a day, 30 mins before meals.
  Interventions: Dietary Supplement: Glucosanol 350mg
- High dose (Glucosanol 500mg) (Experimental): Each capsule contains Glucosanol / Phaselite 500mg
  Subjects will take 2 capsules three times a day, 30 mins before meals.
  Interventions: Dietary Supplement: Glucosanol 500mg

INTERVENTIONS:
Dietary Supplement: Glucosanol 350mg
  Arms: Low dose (Glucosanol 350mg)
Dietary Supplement: Glucosanol 500mg
  Arms: High dose (Glucosanol 500mg)
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
It was proven in a previous clinical study that Glucosanol™ is effective and safe in reducing weight in the overweight and obese. The present study aims at expanding the data concerning the weight management effect of Glucosanol™ in overweight and moderately obese population.

ELIGIBILITY:
Inclusion Criteria:

* BMI 25 kg/m2 - 34,9 kg/m2
* Generally in good health• Desire to lose weight
* Accustomed to regular daily consumption of 3 main meals (breakfast, lunch, dinner)
* Consistent and stable body weight in the last 3 months prior to V1 (less than 5% self-reported change)• Readiness to take IP as recommended
* Readiness to avoid the use of other weight loss and/or management products and/or programs during the study
* Readiness to adhere to diet recommendation during the study
* Readiness to keep the habitual level of physical activity as prior to the study during the study
* Readiness and ability to complete the subject diary and study questionnaires
* Negative pregnancy testing (beta HCG-test in urine) at V1 in women of childbearing potential
* Women of childbearing potential: commitment to use contraception methods

Exclusion Criteria:

* Known allergy or hypersensitivity to the components of the investigational products
* Known allergy or hypersensitivity to members of the Fabaceae family
* Known food allergy (e.g. to cow's milk, eggs, wheat, crustacean, nuts etc.)
* Significant disorders:

  * untreated or unstable thyroid gland disorder
  * untreated or unstable hypertension (>140/90 mm Hg)
  * acute or chronic gastrointestinal (GI) disease or malabsorption disorders (e.g. inflammatory bowel disease, coeliac disease, pancreatitis etc.)
  * diabetes mellitus- coagulation disorder- any other serious organ or systemic diseases that could influence the conduct and/or out-come of the study and/or could affect the tolerability of the subject (in the opinion of the investigator)
* Significant surgery within the last 6 months prior to V1:

  * GI surgery
  * liposuction
* History of eating disorders like bulimia, anorexia nervosa, binge-eating within the last 12 monthsprior to V1
* Clinically relevant excursions of safety laboratoryparameters
* Any electronic medical implant
* Regular use of anticoagulants
* Regular medication and/or supplementation and/or treatment within the last 3 months prior to V1 and during the study:

  * that could influence body weight (e.g. systemic corticosteroids)
  * that could influence gastrointestinal functions (e.g. antibiotics, laxatives, opioids, glucocorticoids, anticholinergics, anti-diarrheals etc.) as per investigator judgement
  * for weight management (e.g. fat binder, carbohydrate/starch blocker, fat burner, satiety products, acupuncture etc.)
* Consumption of food supplements or natural health products for the duration of the study
* Diet to lose and/or manage weight (except ac-cording to the study protocol)
* Vegetarian, vegan or macrobiotic diet
* Smoking cessation within 6 months prior to V1 or during the study (regular smoking during the study at the same level as prior to the study is allowed)
* Pregnancy or nursing
* History of or current abuse of drugs, alcohol or medication
* Inability to comply with study requirements
* Subjects who are deprived of their freedom by administrative or legal decision or who are in guardianship
* Participation in another clinical study in the 30 days prior to V1 and during the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2016-05; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Difference in mean body weight (kg) after 12 weeks of IP intake in comparison between the verum 500mg study arm and placebo | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ralf Uebelhack, MD, Principal Investigator — analyze & realize GmbH
Locations (1):
- Barbara Grube, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jager R, Abou Sawan S, Purpura M, Grube B, Roske Y, De Costa P, Chong PW. Proprietary alpha-amylase inhibitor formulation from white kidney bean (Phaseolus vulgaris L.) promotes weight and fat loss: a 12-week, double-blind, placebo-controlled, randomized trial. Sci Rep. 2024 Jun 3;14(1):12685. doi: 10.1038/s41598-024-63443-8. PMID 38830962